CLINICAL TRIAL: NCT03325972
Title: Randomized, Double-blind, Placebo-controlled Study on the Effects of Intravenous Dexmedetomidine on Pain in Patients Undergoing Elective Spinal Surgery
Brief Title: Study on the Effects of Intravenous Dexmedetomidine on Pain in Patients Undergoing Elective Spinal Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 14-00915
Record Dates: First submitted 2017-10-26; First posted 2017-10-30 (Actual); Results first posted 2023-03-21 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2023-05

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain | interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- IV dexmedetomidine (Experimental): Dexmedetomidine is an alpha-2-adrenergic agonist. It is commonly used for sedation and as an adjunct to general anesthetics.
  Interventions: Drug: Dexmedetomidine
- Placebo (Placebo Comparator): saline placebo
  Interventions: Other: Placebo Saline

INTERVENTIONS:
Drug: Dexmedetomidine — The drug will be administered with a loading dose of 0.5 mcg/kg given over 20 min followed by an infusion at 0.6 mcg/kg/hr. The infusion will be stopped during closure of the fascia.
  Arms: IV dexmedetomidine
Other: Placebo Saline — Placebo will be administered with a loading dose of 0.5 mcg/kg given over 20 min followed by an infusion at 0.6 mcg/kg/hr. The infusion will be stopped during closure of the fascia.
  Arms: Placebo

SUMMARY:
This is a randomized, prospective, double-blind , placebo-controlled trial examining the effects of intraoperative dexmedetomidine infusion on pain in patients undergoing lumbar spinal fusion surgery. One hundred ten subjects (55 in each arm) will be enrolled. Subjects, over the age of 18, undergoing lumbar spinal fusion will be considered eligible for enrollment. Subjects will receive either intraoperative dexmedetomidine or placebo of normal saline infusion. They will be followed for approximately six weeks postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Adults who will undergo lumbar spinal fusion, including surgeries extending into thoracic and sacral segments
* Subject is non-lactating and is either:
* Not of childbearing potential
* Of childbearing potential but is not pregnant at time of surgery as determined by pre-surgical pregnancy testing
* Subject is ASA physical status 1, 2, or 3.

Exclusion Criteria:

* Subject is pregnant or breastfeeding
* Any subject whom the investigators deem unable to complete any/all research related tasks
* Subjects who are cognitively impaired (by history)
* Subject requires antipsychotic medications
* Subject has received treatment with alpha-2 agonists or antagonists within 2 weeks prior to surgery
* Subject has known allergy to dexmedetomidine
* Subjects with impaired renal or hepatic function
* Subjects with advanced heart block
* Subjects with severe ventricular dysfunction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2016-09-14 (Actual); Primary Completion 2022-02-22 (Actual); Study Completion 2022-02-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Doan, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | IV Dexmedetomidine | Placebo
Started | 33 | 31
Completed | 18 | 13
Not Completed | 15 | 18

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IV Dexmedetomidine | Placebo | Total
Number analyzed (Participants) | 33 | 31 | 64
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.2 (8.8) | 59.9 (10.8) | 61.5 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 16 | 35
  Male | 14 | 15 | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 31 | 29 | 60
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 2 | 5
  White | 25 | 27 | 52
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 1 | 4
Region of Enrollment [Number; unit: participants]
  United States | 33 | 31 | 64

OUTCOME MEASURES:

1. Primary Outcome: Morphine Equivalents Used During the First 48 Hours Post-Surgery
Description: Amount of morphine administered during the 48 hours following surgery.
Time Frame: Up to 48 Hours Post-Surgery (Day 2)
Measure: Median (Inter-Quartile Range); unit: morphine milligram equivalent (MME)
Arm/Group | IV Dexmedetomidine | Placebo
Number analyzed (Participants) | 33 | 30
morphine milligram equivalent (MME) | 180 [120 to 309.5] | 142.5 [76.5 to 211.5]

2. Secondary Outcome: Mean Numeric Pain Rating Scale (NRS) Scores During the First 48 Hours Post-Surgery
Description: The NPRS is a self-assessment of pain. Participants select a number between 0 and 10 that fits best to their pain intensity, where 0 represents 'no pain at all' and 10 represents 'the worst pain ever possible.'
Time Frame: 48 Hours Post-Surgery (Day 2)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IV Dexmedetomidine | Placebo
Number analyzed (Participants) | 32 | 30
score on a scale | 7.27 (1.96) | 6.53 (2.12)

3. Secondary Outcome: Numeric Pain Rating Scale (NPRS) Score at 6 Weeks Post-Surgery
Description: as for outcome 2
Time Frame: Week 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IV Dexmedetomidine | Placebo
Number analyzed (Participants) | 26 | 19
score on a scale | 3 (2.61) | 3.26 (2.53)

4. Secondary Outcome: Morphine Equivalents Used at 6 Weeks Post-Surgery
Description: Amount of morphine administered during the 6 weeks following surgery.
Time Frame: Up to Week 6
Measure: Median (Inter-Quartile Range); unit: morphine milligram equivalent (MME)
Arm/Group | IV Dexmedetomidine | Placebo
Number analyzed (Participants) | 22 | 18
morphine milligram equivalent (MME) | 0 [0 to 6.25] | 0 [0 to 1.25]

5. Secondary Outcome: Number of Participants Requiring Pressor Use During Intraoperative Period
Description: The intraoperative period begins when the patient is transferred to the operating room table and ends with the transfer of a patient to the Post Anesthesia Care Unit (PACU).
Time Frame: From beginning up to end of surgery (Day 0 - typically 1 to 3 hours)
Measure: Count of Participants; unit: Participants
Arm/Group | IV Dexmedetomidine | Placebo
Number analyzed (Participants) | 33 | 31
Participants | 25 | 20

6. Secondary Outcome: Number of Participants Requiring Pressor Use During First 48-Hours Post-Surgery
Time Frame: Up to 48 Hours Post-Surgery (Day 2)
Measure: Count of Participants; unit: Participants
Arm/Group | IV Dexmedetomidine | Placebo
Number analyzed (Participants) | 33 | 30
Participants | 7 | 2

7. Secondary Outcome: Length of PACU Stay
Time Frame: From PACU admission up to end of PACU stay (Day 0 - typically 1 to 3 hours)
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | IV Dexmedetomidine | Placebo
Number analyzed (Participants) | 32 | 30
minutes | 172 (90.24) | 152 (58.77)

8. Secondary Outcome: Length of Hospital Stay
Time Frame: From admission up to discharge (Up to 6 Weeks)
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | IV Dexmedetomidine | Placebo
Number analyzed (Participants) | 33 | 31
Days | 5.89 (2.55) | 5.03 (2.42)

9. Secondary Outcome: Mean Quality of Recovery After Anesthesia (QoR-15) Scores During the First 48 Hours Post-Surgery
Description: The QoR-15 is a 15-item self measurement of patients' overall satisfaction with postoperative recovery. Items are ranked on a Likert scale of 0 to 10, where: 0 = none of the time [poor] and 10 = all of the time [excellent]. Higher scores indicate greater satisfaction with postoperative recovery. The total score ranges from 0 to 150; higher scores indicate greater satisfaction with postoperative recovery.
Time Frame: 48 Hours Post-Surgery (Day 2)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IV Dexmedetomidine | Placebo
Number analyzed (Participants) | 32 | 30
score on a scale | 90.73 (16.72) | 89.3 (21.03)

10. Secondary Outcome: Quality of Recovery After Anesthesia (QoR-15) Score at 6 Weeks Post-Surgery
Description: as for outcome 9
Time Frame: Week 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IV Dexmedetomidine | Placebo
Number analyzed (Participants) | 24 | 18
score on a scale | 115.5 (16.91) | 120.67 (16.57)

11. Secondary Outcome: Mean Short-Form McGill Pain Questionnaire (SF-MPQ) Scores During First 48 Hours Post-Surgery
Description: The SF-MPQ is a self-assessment of pain symptoms. The questionnaire includes 15 pain descriptor items that are ranked on a Likert scale from 0 (none) to 3 (severe); one Visual Analogue Scale (VAS) item on which participants rank pain on a 10 cm VAS; and one Present Pain Intensity item on which participants rank their present pain on a Likert scale from 0 (no pain) to 5 (excruciating). The total score is the sum of responses and ranges from 0-60; lower scores indicate less pain. The SF-MPQ is administered on postoperative days 1 and 2.
Time Frame: 48 Hours Post-Surgery (Day 2)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IV Dexmedetomidine | Placebo
Number analyzed (Participants) | 31 | 30
score on a scale | 27.9 (8.9) | 25.5 (10.7)

12. Secondary Outcome: Short-Form McGill Pain Questionnaire (SF-MPQ) Scores at 6 Weeks Post-Surgery
Description: The SF-MPQ is a self-assessment of pain symptoms. The questionnaire includes 15 pain descriptor items that are ranked on a Likert scale from 0 (none) to 3 (severe); one Visual Analogue Scale item on which participants rank pain on a 10 cm VAS; and one Present Pain Intensity item on which participants rank their present pain on a Likert scale from 0 (no pain) to 5 (excruciating). The total score is the sum of responses and ranges from 0-60; lower scores indicate less pain.
Time Frame: Week 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IV Dexmedetomidine | Placebo
Number analyzed (Participants) | 26 | 19
score on a scale | 15.2 (23.1) | 12.2 (11.4)

ADVERSE EVENTS:
Time Frame: 6 weeks following last administration of study treatment
Description: At each contact with the participant, the investigator requested information on adverse events by specific questioning and, as appropriate, by examination.
Arm/Group | IV Dexmedetomidine | Placebo
All-Cause Mortality (participants affected / at risk) | 1/33 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/31
Other Adverse Events (participants affected / at risk) | 1/33 | 2/31
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | IV Dexmedetomidine (N=33) | Placebo (N=31)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Bradycardia (Cardiac disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-27): https://cdn.clinicaltrials.gov/large-docs/72/NCT03325972/Prot_SAP_000.pdf